CLINICAL TRIAL: NCT05920148
Title: The Effect of Total Knee Replacement Surgery on Immune Functioning in Elderly
Brief Title: The Immu-KNEE-ty Study
Status: Completed | Type: Observational
Sponsor: Wageningen University (Other)
Collaborators: Wageningen University and Research (Other); Gelderse Vallei Hospital (Other)
Responsible Party: Principal Investigator, Klaske van Norren, Principle Investigator / Associate Professor, Wageningen University
Other Study IDs: NL84069.091.23
Record Dates: First submitted 2023-06-15; First posted 2023-06-27 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-06

CONDITIONS: Immunosenescence; Aging
Keywords: Knee arthroplasty; Elderly; Immune functioning; Monocytes
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Elderly
  Interventions: Procedure: Knee arthroplasty

INTERVENTIONS:
Procedure: Knee arthroplasty — At multiple timepoints (i.e., ± 6 weeks before, and 1 day, 1 week, ± 2 weeks, and ± 6 weeks after surgery) before and after total knee replacement surgery blood will be collected to assess immune functioning

SUMMARY:
The goal of this observational study is to determine changes in immune functioning after total knee replacement surgery in elderly. The study population consists of 14 patients aged 65 years or over undergoing primary total knee replacement surgery. Immune functioning will be assessed at multiple timepoints before and after surgery (i.e., ± 6 weeks before, and 1 day, 1 week, ± 2 weeks, and ± 6 weeks after surgery). Each patient will serve as his/her own control. Immune functioning will primarily be assessed by determining the change from baseline in monocyte-derived TNFα production at 1 week after surgery. Changes in monocyte responsiveness are considered indicative for changes in immune functioning. As secondary objective, additional parameters of immune functioning will be assessed. In addition, the course of immune functioning following total knee replacement surgery will be investigated. Burden and potential risks for the patient are estimated to be minor. During the study, 5 blood samples of 20 mL will be collected over a period of ± 12 weeks, resulting in a total blood draw of 100 mL. During surgery a sample of synovial fluid (± 2 mL) will be taken from surgical waste. Before and after surgery patients will report their pain medication intake and the presence of cold and flu-like symptoms in a diary. Patients do not directly benefit from the study.

DETAILED DESCRIPTION:
The world population is progressively aging. As humans age, their immune system becomes weaker through a process called immunosenescence. This age-related decline in immune functioning results in an increased susceptibility to infections. Elderly with chronic diseases or elderly who have experienced an incident, such as fall-related trauma or surgery, are particularly vulnerable to these infections, likely due to immunosuppression resulting from such an immune challenge. Currently, there are no standard interventions used to improve immune functioning in these immune-suppressed elderly. However, before the potential of such interventions can be explored, postoperative immune suppression in elderly first needs to be demonstrated.

The goal of this prospective ex vivo study is therefore to determine changes in immune functioning after total knee replacement surgery in elderly.

The study population consists of 14 patients (classified as ASA II or ASA III) aged 65 years or over, diagnosed with osteoarthritis, undergoing primary total knee replacement surgery under general anesthesia.

Immune functioning will be assessed at multiple timepoints before and after surgery (i.e., ± 6 weeks before, and 1 day, 1 week, ± 2 weeks, and ± 6 weeks after surgery). Each patient will serve as his/her own control. Immune functioning will primarily be assessed by determining the change from baseline in monocyte-derived TNFα production at 1 week after surgery. TNFα production will be measured after ex vivo stimulation of whole blood with inflammatory stimuli and normalized for monocyte count. Changes in monocyte responsiveness are considered indicative for changes in immune functioning.

As secondary objective, additional parameters of immune functioning will be assessed. In addition, the course of immune functioning following total knee replacement surgery will be investigated.

Burden and potential risks for the patient are estimated to be minor. During the study, 5 blood samples of 20 mL will be collected over a period of ± 12 weeks, resulting in a total blood draw of 100 mL. Blood sampling will be combined with regular care visits, with the exception of one occasion where blood sampling will be performed at home. Patients could experience mild pain by the venipuncture, which occasionally leads to lightheadedness, fainting and hematoma. During surgery a sample of synovial fluid (± 2 mL) will be taken from surgical waste. Before and after surgery patients will report their pain medication intake and the presence of cold and flu-like symptoms in a diary. Patients do not directly benefit from the study.

ELIGIBILITY:
Inclusion Criteria:

* Planned for primary total knee replacement surgery
* Aged 65 years or over
* Diagnosed with osteoarthritis
* ASA Physical Status Classification of II or III
* Willing to donate a blood sample at 5 different timepoints
* Able to give written informed consent

Exclusion Criteria:

* Daily use of high doses NSAIDs within the 14 days before inclusion: Defined as higher than maintenance dose in the "farmacotherapeutisch kompas". For example: acetylsalicylic acid > 4 g/day; diclofenac > 75 mg/day; naproxen > 500 mg/day; ibuprofen> 1600 mg/day; celecoxib > 200 mg/day
* Use of systemic corticosteroids
* Use of antibiotics within the 14 days before inclusion
* Current diagnosis of cancer
* Diagnosed with a primary immunodeficiency disorder (e.g., Severe Combined Immunodeficiency (SCID), Common Variable Immune Deficiency (CVID), X-linked agammaglobulinemia, selective immunoglobulin A deficiency, chronic granulomatous disease)
* Vaccination (e.g., immunization against COVID-19, influenza, pneumonia, and travel-related infections) within the 14 days before inclusion and during the study period
* Current participation in other scientific research

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consists of 14 patients (classified as ASA II or ASA III) aged 65 years or over, diagnosed with osteoarthritis, undergoing primary total knee replacement surgery.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Monocyte-derived TNFa production | Change from baseline at 1 week after surgery
  TNFα production after ex vivo stimulation of whole blood with inflammatory stimuli corrected for monocyte count

SECONDARY OUTCOMES:
Monocyte-derived cytokine production | Change from baseline at 1 day after surgery
  Cytokine production after ex vivo stimulation of whole blood with inflammatory stimuli and corrected for monocyte count
Monocyte-derived cytokine production | Change from baseline at 1 week after surgery
  Cytokine production after ex vivo stimulation of whole blood with inflammatory stimuli and corrected for monocyte count
Monocyte-derived cytokine production | Change from baseline at ± 2 weeks after surgery
  Cytokine production after ex vivo stimulation of whole blood with inflammatory stimuli and corrected for monocyte count
Monocyte-derived cytokine production | Change from baseline at ± 6 weeks after surgery
  Cytokine production after ex vivo stimulation of whole blood with inflammatory stimuli and corrected for monocyte count
Monocyte-derived cytokine production | Change from baseline at 1 day after surgery
  Cytokine production after ex vivo stimulation of isolated monocytes with inflammatory stimuli
Monocyte-derived cytokine production | Change from baseline at 1 week after surgery
  Cytokine production after ex vivo stimulation of isolated monocytes with inflammatory stimuli
Monocyte-derived cytokine production | Change from baseline at ± 2 weeks after surgery
  Cytokine production after ex vivo stimulation of isolated monocytes with inflammatory stimuli
Monocyte-derived cytokine production | Change from baseline at ± 6 weeks after surgery
  Cytokine production after ex vivo stimulation of isolated monocytes with inflammatory stimuli
PBMC (peripheral blood mononuclear cell)-derived cytokine production | Change from baseline at 1 day after surgery
  Cytokine production after ex vivo stimulation of PBMCs with inflammatory stimuli
PBMC-derived cytokine production | Change from baseline at 1 week after surgery
  Cytokine production after ex vivo stimulation of PBMCs with inflammatory stimuli
PBMC-derived cytokine production | Change from baseline at ± 2 weeks after surgery
  Cytokine production after ex vivo stimulation of PBMCs with inflammatory stimuli
PBMC-derived cytokine production | Change from baseline at ± 6 weeks after surgery
  Cytokine production after ex vivo stimulation of PBMCs with inflammatory stimuli
Composition of immune cell populations | Change from baseline at 1 day after surgery
  Composition of immune cell populations (white blood cell count and differential) in whole blood
Composition of immune cell populations | Change from baseline at 1 week after surgery
  Composition of immune cell populations (white blood cell count and differential) in whole blood
Composition of immune cell populations | Change from baseline at ± 2 weeks after surgery
  Composition of immune cell populations (white blood cell count and differential) in whole blood
Composition of immune cell populations | Change from baseline at ± 6 weeks after surgery
  Composition of immune cell populations (white blood cell count and differential) in whole blood
Systemic inflammation | Change from baseline at 1 day after surgery
  Systemic inflammation as measured by circulating cytokines, chemokines, acute phase proteins, oxylipins, and markers of intestinal function
Systemic inflammation | Change from baseline at 1 week after surgery
  Systemic inflammation as measured by circulating cytokines, chemokines, acute phase proteins, oxylipins, and markers of intestinal function
Systemic inflammation | Change from baseline at ± 2 weeks after surgery
  Systemic inflammation as measured by circulating cytokines, chemokines, acute phase proteins, oxylipins, and markers of intestinal function
Systemic inflammation | Change from baseline at ± 6 weeks after surgery
  Systemic inflammation as measured by circulating cytokines, chemokines, acute phase proteins, oxylipins, and markers of intestinal function
Phagocytic function of monocytes | Change from baseline at 1 day after surgery
  Phagocytic function of monocytes as measured by the uptake of fluorescent particles
Phagocytic function of monocytes | Change from baseline at 1 week after surgery
  Phagocytic function of monocytes as measured by the uptake of fluorescent particles
Phagocytic function of monocytes | Change from baseline at ± 2 weeks after surgery
  Phagocytic function of monocytes as measured by the uptake of fluorescent particles
Phagocytic function of monocytes | Change from baseline at ± 6 weeks after surgery
  Phagocytic function of monocytes as measured by the uptake of fluorescent particles
Monocyte HLA-DR expression | Change from baseline at 1 day after surgery
  Monocyte HLA-DR expression as measured with fluorescent antibodies
Monocyte HLA-DR expression | Change from baseline at 1 week after surgery
  Monocyte HLA-DR expression as measured with fluorescent antibodies
Monocyte HLA-DR expression | Change from baseline at ± 2 weeks after surgery
  Monocyte HLA-DR expression as measured with fluorescent antibodies
Monocyte HLA-DR expression | Change from baseline at ± 6 weeks after surgery
  Monocyte HLA-DR expression as measured with fluorescent antibodies
Synovial inflammation | During surgery
  Synovial inflammation as scored by the surgeon (yes/no)
Synovial inflammation | During surgery
  Synovial inflammation as measured by cytokine and chemokine levels in synovial fluid

OTHER OUTCOMES:
Body Mass Index | Baseline
  Body Mass Index
American Society of Anesthesiologists (ASA) classification | Baseline
  ASA classification
Kellgren-Lawrence classification | Baseline
  Kellgren-Lawrence classification
Knee function and pain | Baseline
  Knee function and pain as measured by the Oxford Knee Score (OKS)
Physical function | Baseline
  Physical function as measure by the Knee injury and Osteoarthritis Outcome Score - Physical Function Short Form (KOOS-PS)
Quality of Life (QoL) | Baseline
  QoL as measured by EQ-5D
Pain as measured by the Numeric Pain Rating Scale (NPRS) | Baseline
  Pain as measured by the NPRS
Mobility | Baseline
  Timed Up and Go (TUG) test
Mobility | Baseline
  Sit to Stand (STS) test
Mobility | Baseline
  10 Meter Walk Test (10MWT)
Duration of surgery | During surgery
  Duration of surgery
Amount of blood loss | During surgery
  Amount of blood loss
Analgesic therapies | 1 week before surgery
  Amount of analgesic therapies recorded in a pain medication diary
Analgesic therapies | During hospitalization
  Amount of analgesic therapies recorded in a pain medication diary
Analgesic therapies | In the 6 weeks after surgery
  Amount of analgesic therapies recorded in a pain medication diary
Cold and flu-like symptoms | In the 6 weeks after surgery
  Cold and flu-like symptoms in a diary

CONTACTS AND LOCATIONS:
Locations (1):
- Gelderse Vallei Hospital, Ede, Netherlands

IPD SHARING:
Plan to Share IPD: No